CLINICAL TRIAL: NCT04772872
Title: NEURODEVELOPMENTAL OUTCOMES OF SINGLETON CONCEIVED FROM FRESH AND FROZEN EMBRYO TRANSFER COMPARED WITH NATURALLY CONCEIVED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sally Ashraf Mohammed Askar, Principle investigator, Cairo University
Other Study IDs: Sasker_phd2021
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Singeleton Conceived Fresh and Frozen Embryo Transfer (ICSI/IVF), Naturally Conceived

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A:Naturally conceived singleton: * Neonatal neurobehavior will be measured by Brazelton neonatal behavior assessment scale.
  * Neonatal maturity will be represented by the variance of estimated gestational age that determined by new Ballard score.
  * Apgar score will be represented by the variance of degree of scores.
  * Birth weight will be measured in grams.
  Interventions: Other: Assessment by Brazelton neonatal behavior for group A,Band C
- Group B: Singleton conceived from fresh embryo transfer(IVF/ICSI): * Neonatal neurobehavior will be measured by Brazelton neonatal behavior assessment scale.
  * Neonatal maturity will be represented by the variance of estimated gestational age that determined by new Ballard score.
  * Apgar score will be represented by the variance of degree of scores.
  * Birth weight will be measured in grams.
  Interventions: Other: Assessment by Brazelton neonatal behavior for group A,Band C
- Group C: Singleton conceived from frozen embryo transfer (IVF/ICSI): * Neonatal neurobehavior will be measured by Brazelton neonatal behavior assessment scale.
  * Neonatal maturity will be represented by the variance of estimated gestational age that determined by new Ballard score.
  * Apgar score will be represented by the variance of degree of scores.
  * Birth weight will be measured in grams.
  Interventions: Other: Assessment by Brazelton neonatal behavior for group A,Band C

INTERVENTIONS:
Other: Assessment by Brazelton neonatal behavior for group A,Band C — * Neonatal neurobehavior will be measured by Brazelton neonatal behavior assessment scale.
  * Neonatal maturity will be represented by the variance of estimated gestational age that determined by new Ballard score.
  * Apgar score will be represented by the variance of degree of scores.
  * Birth weight will be measured in grams.
  Other Names: Assessment by new ballard score for group A,Band C; Assessment infant weight scale for group A,Band C; assessment by APGAR score for group A,B and C

SUMMARY:
This study aimed to: detect difference in neurobehavior, maturity, Apgar score and birth weight of singleton conceived from fresh and frozen embryo transfer and naturally conceived.

DETAILED DESCRIPTION:
The use of ART has increased significantly during the past decades with more than 390000 children born worldwide annually and the total number of ART children now exceeding 7 million (Adamson et al., 2018). ART is associated with an increased risk of perinatal complications, including preterm birth (PTB) and small for gestational age (SGA) (Pandey et al., 2012 and Pinborg et al., 2013).

When mothers had been received ovarian stimulation in ART, multiple follicles and corpora lutea are produced, which produce supraphysiologic serum levels of multiple hormones and other factors, including estradiol, progesterone, and vascular endothelial growth factor (VEGF). This non physiological hormonal milieu affects both the endometrium and the embryo, potentially resulting in altered growth of the developing fetus. There was a serious effect of the supraphysiologic hormonal environment on pregnancy outcomes. (Imudia et al., 2012).

Neonates born after an IVF/ICSI procedure have an increased risk of various developmental problems, neurological disabilities, impairments or handicap, especially the cerebral palsy (CP) (Strömberg et al., 2002 and Squires and Kaplan, 2007).The increased risk of prematurity and smaller birth weight after an ART procedure required regular periodic screening and careful developmental follow-up of these children. (Boulet et al., 2008).

Singleton born after an IVF procedure were more likely to need habilitation treatment and had increased risk of developing neurological problems, especially cerebral palsy (CP), suspicion for a delay in their development. (Strömberg et al., 2002) Children born after an IVF procedure had three times higher presence of CP compared to the children from the general population and the risk of suspicion for a delay in their development was four times higher in children born after an IVF procedure than in the naturally conceived. (Strömberg et al., 2002). There is evidence of associations among the ART procedure and the developmental delay (Hvidtjørn et al., 2009).

The lack of early examination of neonates׳s neurobehavior conceived from ICSI/IVF may be led to developmental delay in these neonates. Early detection of neurobehavior deviation is essential for effective control of this potentially debilitating morbidity. As there is no available data about neurobehavior of Egyptian neonates conceived from frozen and fresh embryo transfer so there is an arising need to address this gap of knowledge.

Thus, to overcome previous limitation, the current study aimed to evaluate neurobehavior of singletons conceived from fresh and frozen embryo transfer compared with naturally conceived and screening for identify need for early intervention and developmental follow up to prevent worsening and progression of dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

* Singleton born through IVF/ICSI (frozen embryo transfer and fresh embryo transfer) after 37 weeks of gestation.
* Singleton whose mothers are aged from 25 to 35 years old and has BMI ranged from 18.5 to 29.

Exclusion Criteria:

* Singleton will be excluded from study if one or more of the following is present:

  1. vanishing twins (singleton birth where a twin pregnancy recorded at 7 weeks of gestational age (double heart rate at sound)).
  2. Preterm singleton.
  3. Congenital anomalies
  4. Gestational surrogates.
  5. Donor oocyte pregnant.
  6. Multiple birth.
  7. Singleton whose mothers have

     * Metabolic diseases (hypertension and diabetes).
     * Chronic health issues (asthma and epilepsy).
     * Gestational condition (preeclampsia, impaired glucose tolerance, gestational diabetes, anemia and ULT occurrence).
     * Placenta previa and placenta accrete.
     * Premature rapture of membrane.
     * Premature uterine contraction.
     * Cervical insufficiency.
     * Smoker mother.

Ages: 1 Hour to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 186 full term singletons born through IVF/ICSI after 37 weeks of gestation and from naturally conceived will be enrolled in this study
Sampling Method: Probability Sample
Enrollment: 186 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Neurobehavior | at first day of birth
  Brazelton behavioral neonatal assessment (BNBAS) The NBAS assesses the infant's behavioral capacities, including his or her ability to respond to the environment, such as the ability to orient and habituate to visual or auditory stimuli, both animate and inanimate; the quality of motor tone and activity levels elected priories those that potentially reflect skills associated with attention
maturity | at first day of birth
  New Ballard Score New Ballard score was rapid, accurate method of clinically assessing gestational maturation of newly born infants developed by Dr. Jeanne L Ballard. (Ballard et al., 1991).
  The New Ballard Score is a set of procedures to determine Gestational age through neuromuscular and physical assessment of a newborn infant.:
  * Neuromuscular maturity contains: posture, square window, assessing the flexibility of the wrist, arm recoil, popliteal angle, scarf sign and heel to ear.
  * The physical assessment contains: skin, ear/eye, lanugo hair, plantar surface, breast bud and genitals. (Appendix III) This scoring used for the estimation of age in the range of 26 gestational weeks to 44 gestational weeks.
birth weight | at first day of birth
  Weight record is essential to monitor the adequacy of nutrition as well as fluid balance. Weight of birth is the single most useful predictor of neonatal morbidity and mortality. A weighing scale for measuring the weight at birth is essential for all facilities where deliveries take place and where neonates are looked after
Apgar scoring | at first day of birth
  Apgar scoring The Apgar score, the first test given to new born, assessed in the delivery or birthing room after the fetus birth. The test was designed to quickly evaluate a newborn's physical condition and to see if there is an immediate need for extra medical or emergency care. It was done at 1 minute and 5 minutes after birth, newborns are observed and rated according to the Apgar score

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided